CLINICAL TRIAL: NCT03444779
Title: Comparative Evaluation of Minimally Invasive "tibial Tuberoplasty" Surgical Technique Versus Conventional Open Surgery for Tibial Plateau Fractures (TUBERIMPACT Study)
Brief Title: Comparative Evaluation of Minimally Invasive "tibial Tuberoplasty" Surgical Technique Versus Conventional Open Surgery for Tibial Plateau Fractures
Acronym: TUBERIMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A01027-48
Record Dates: First submitted 2018-02-02; First posted 2018-02-23 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Schatzker Type 2 or 3 Tibial Plateau Fracture
Keywords: tibial plateau fracture; minimally invasive surgery; ballon reduction
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Open Abdomen Techniques

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient blinded until D2 visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): The patients will be treated with an open technique: cutaneous incision with submeniscal arthrotomy under guidance of a fluoroscope. The reduction will be performed using a spatula, a bone tamp or open reduction internal fixation. The osteosynthesis and filling of the cavity will be performed by the same surgical access.
  Interventions: Device: Open technique
- Experimental group (Experimental): The patients will be treated with the "Tibial Tuberoplasty" technique under fluoroscopic guidance with or without arthroscopy. The reduction will be performed by an anterior approach using a kyphoplasty balloon. The combined osteosynthesis including cannulated screws and cementoplasty will both be performed by a percutaneous technique.
  Interventions: Device: Tibial Tuberoplasty

INTERVENTIONS:
Device: Tibial Tuberoplasty — Kyphoplasty ballon
  Arms: Experimental group
Device: Open technique — Cutaneous incision with submeniscal arthrotomy under guidance of a fluoroscope.
  Arms: Control group

SUMMARY:
PMSI (French Medico-Administrative Database) data shows more than 10000 proximal tibial fractures diagnosed in 2014 and 4055 lateral tibial plateau fractures operated in 2013 in France. 50% of these surgical fractures is related to the lateral condyle and causes split/depression (Schatzker 2) or pure depression (Schatzker 3). This high rate results from the recent democratization of high-risk sports, as well as an aging population with increased risks of falling. Aside from the resulting reduced physical activity, the social and professional impact of these fractures is undeniable and represents significant costs for our health care system. A recently published prospective case series reports 28 job losses out of 41 patients treated.

The clinical outcome of these patients depends mainly on the primary stability provided by the surgical treatment, after the greatest anatomical reduction possible. Indeed, Giannoudis and al. have demonstrated that under simple X-rays, the smaller the detected step-off, the better the outcome.The aim is to allow for recovery of good joint mobility to promote rapid resumption of activity and to limit the onset of early osteoarthritis.

The classical technique used for reduction and osteosynthesis of tibial plateau fractures (open surgical technique using a bone tamp) has several pitfalls : devascularization of the bone and skin, risks of infection and functional rehabilitation difficulties with delayed recovery of weight bearing. Moreover, this technique does not allow for the simultaneous diagnosis and treatment of other possible lesions, such as meniscal injuries in particular.

Since 2011, Poitiers University Hospital is offering to its patients a new minimally invasive technique for the reduction and stabilization of tibial plateau fractures, baptized "Tibial Tuberoplasty". The concept derives from the divergent use of vertebral kyphoplasty, initially dedicated for spinal injuries and transposed here to the tibial plateau. This technique involves expansion of the tibial plateau through inflation of a kyphoplasty balloon, filling of the created cavity with cement (PMMA, calcium phosphate) and percutaneous screw fixation.

Orthopaedic surgeons of Poitiers University Hospital performed the first tibial tuberoplasties through a feasibility study on 36 cadaveric subjects and then transposed the technique to human. Surgeons identified major advantages such as minimal skin damage, possible treatment of posterior and multi-fragmented compressions (lifting in a single block by the balloon), reinforcement of the stability of the assembly using cement, possible use of combined arthroscopy (for concomitant meniscal injuries treatment).

This technique allows for optimization of the fracture reduction by elevating the posterior fragments with the inflatable bone tamp through an anterior approach. The reduction is made possible thanks to the specificity of the inflatable bone tamp which inflates and reduces the area of least resistance.

The aim of this innovative technique is focused on the anatomical reduction in order to restore the convexity of the tibial plateau which is similar to the balloon convexity.

The results from the first 40 patients operated since 2011 are promising and show a proportion of 70% presenting less than 5 mm step-off reduction. A larger scale multicenter randomized controlled trial is now requested to further demonstrate the superiority of the "Tibial Tuberoplasty" to the standard treatment.

The coordinator investigator designed this study to evaluate the quality of tibial fracture reduction offered by percutaneous "Tibial Tuberoplasty" versus conventional open surgery for tibial plateau fracture but also its impact on clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patients with a Schatzker type 2 or 3 tibial plateau fracture (compression with or without split) demonstrated on CT-scan and located in the lateral or medial condyle of tibia.
3. Patients with fractures caused by trauma.
4. Patients with fractures 10 days old maximum.
5. Understand and accept the constraints of the study.
6. Be a beneficiary or affiliated member of a Health Insurance plan.
7. Give written consent for the study after having received clear information.

Exclusion Criteria:

1. Age < 18 years old.
2. Patients with fractures resulting from osteolysis.
3. Patients with open fractures.
4. Patients with fractures more than 10 days old.
5. Patients with concomitant fracture(s) or condition(s) during the trauma reducing the range of motion.
6. Patients unable to walk before the injury.
7. History of sepsis in the injured knee.
8. Contraindications to anesthesia, contrast agent, medical devices or cement.
9. History of hypersensitivity reactions to contrast media, bone filler or metal.
10. Patients with a degenerative joint disease (polyarthritis, etc.).
11. Absence of signature of the informed consent form.
12. Patients not covered by French national health insurance.
13. Subjects requiring closer protection, i.e. minors, pregnant women, nursing mothers, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection, and finally patients in an emergency setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Post-operative radiological step-off reduction blindly measured by high resolution CT-scan | Day 2
  Compare step-off anatomical reduction of tibial plateau fracture by "Tibial Tuberoplasty" versus conventional open surgery using CT-scan

SECONDARY OUTCOMES:
Knee range of motion (degrees) | Day 21, Day 45, Month 3, Month 6, Month 12 and Month 24
  Knee range of motion
Numeric Pain Rating Scale | Inclusion, Day 2, Day 21, Day 45, Month 3, Month 6, Month 12 and Month 24
  The NPRS is an 11-point scale from 0-10 ("0" = no pain and "10" = the most intense pain imaginable). Patients verbally select a value that is most in line with the intensity of pain that they have experienced in the last 24 hours.
Knee injury and Osteoarthritis Outcome Score | Inclusion, Day 21, Day 45, Month 3, Month 6, Month 12 and Month 24
  The KOOS questionnaire is a functional score validated in the French language and one of the only validated in knee trauma. The Knee injury and Osteoarthritis Outcome Score (KOOS) was developed as an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis. The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). The KOOS has been validated for several orthopaedic interventions such as anterior cruciate ligament reconstruction, meniscectomy and total knee replacement.
Score on Euro Quality of Life-5 Dimension Health questionnaire | Inclusion, Day 45, Month 3, Month 6, Month 12 and Month 24
  The EQ-5D-5L is a standardized instrument used to measure health-related quality of life (HRQoL) which comprises a descriptive system and a visual analogue scale. The descriptive system is composed of 5 questions assessing mobility, self-care, usual activities, pain/discomfort and anxiety/depression with 5 possible responses for each item: 1- no problems, 2- slight problems, 3- moderate problems, 4- severe problems and 5- extreme problems). A global index with a maximum score of 1 is calculated from the responses to these 5 dimensions by means of normograms. The maximum score of 1 indicates the best possible quality of life. The visual analogue scale ranging from 0 to 100 also allows the patient to rate his/her perceived quality of life, where 100 indicates the best possible quality of life.
Description of Adverse events | from Inclusion to Month 24 (End Of Study)
  Adverse events
Time to partial and full weight-bearing | from Day 0 (surgery) to Month 24 (End Of Study)
  Time to partial and full weight-bearing

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy VENDEUVRE, Dr, Principal Investigator — Poitiers Hospital University
Locations (12):
- France (11):
  - CHU d'Amiens, Amiens
  - CHU Angers, Angers
  - AP-HP / Hopital Ambroise Paré, Boulogne-Billancourt
  - CHU de Brest, Brest
  - CHU Dijon, Dijon
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU Rouen, Rouen
  - CHRU Tours, Tours
  - CH Versailles, Versailles
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vendeuvre T, Monlezun O, Brandet C, Ingrand P, Durand-Zaleski I, Gayet LE, Germaneau A, Khiami F, Roulaud M, Herpe G, Rigoard P. Comparative evaluation of minimally invasive 'tibial tuberoplasty' surgical technique versus conventional open surgery for Schatzker II-III tibial plateau fractures: design of a multicentre, randomised, controlled and blinded trial (TUBERIMPACT study). BMJ Open. 2019 Sep 3;9(8):e026962. doi: 10.1136/bmjopen-2018-026962. PMID 31481365